CLINICAL TRIAL: NCT00004804
Title: Phase III Randomized Study of High Vs Standard Dose of Interferon Alfa for Chronic Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Tulane University School of Medicine (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11964; TUMC-M1260
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-02

CONDITIONS: Hepatitis C
Keywords: hepatitis C; immunologic disorders and infectious disorders; rare disease; viral infection
MeSH Terms: conditions — Hepatitis C; Immune System Diseases; Communicable Diseases; Rare Diseases; Virus Diseases | interventions — Interferon-alpha

INTERVENTIONS:
Drug: interferon alfa

SUMMARY:
OBJECTIVES: I. Determine whether the initial response to interferon alfa (IFN-A) can be increased by starting at a dose of 5 MU three times a week in patients with chronic hepatitis C.

II. Determine whether patients who had normalized alanine aminotransferase (ALT) levels can maintain normal ALT during stepwise dose reduction from 5 MU to 3 MU to 1.5 MU.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are randomly assigned to 1 of 2 treatment groups in a 2:1 ratio.

The first group is treated with high-dose interferon alfa (IFN-A) administered subcutaneously twice a week for 12 weeks. If the alanine aminotransferase (ALT) level has normalized, the IFN-A dose is decreased in a stepwise fashion. If the ALT level decreases by more than 50%, IFN-A is continued at the same dose until week 24 or the ALT normalizes. If the ALT level decreases by less than 50%, treatment is discontinued.

The second group is treated with standard-dose IFN-A administered subcutaneously twice a week for 24 weeks.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Biopsy-proven chronic hepatitis Anti-hepatitis C virus positive Hepatitis B surface antigen negative
* No decompensated cirrhosis

--Prior/Concurrent Therapy--

* No concurrent immunosuppressives At least 1 year since interferon

--Patient Characteristics--

* Hepatic: No other cause of liver disease
* Other: Not HIV positive

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57
Dates: Start 1993-08

CONTACTS AND LOCATIONS:
Overall Officials: Anna S. F. Lok, Study Chair — Tulane University School of Medicine